CLINICAL TRIAL: NCT04860349
Title: Effects of High Intensity Interval Training on Waist Circumference and Fat Percentage at Trunk Region Among Physically Inactive Overweight Young Adults
Brief Title: Is High Intensity Interval Training Effective to Reduce the Waist Circumference and Fat Percentage at Trunk Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Principal Investigator, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U/SERC/92/2021
Record Dates: First submitted 2021-04-16; First posted 2021-04-26 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Overweight; Physically Inactive; Adults
MeSH Terms: conditions — Overweight | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (Experimental): 20 minutes of High Intensity Interval Training for experimental group.
  Interventions: Other: High Intensity Interval Training
- Control (No Intervention): No intervention for the control group.

INTERVENTIONS:
Other: High Intensity Interval Training — 4-weeks of high intensity interval training, 3 sessions/week on alternate days. each session for 20 minutes, excluding the warm-up and cool-down.
  Arms: High Intensity Interval Training

SUMMARY:
Overweight is a risk factor for a number of non-communicable diseases, and this risk doubles, if an individual is physically inactive. Various exercise interventional protocols in the past have been reported on treating overweight and obesity which helps to decrease the different anthropometric variables. Despite all these protocols, obese and overweight do not seem to benefit greatly by these exercise training programs, as lack of time is thought to the main reason for not engaging in healthful physical exercise. Research evidence has proven that people with a body mass index of more than 30 kg/m2 and waist circumference of more than 102 cm have 2-fold higher risk of waking fewer steps daily. Although physical exercise is thought to be very helpful in regulating the body weight, it is very important to identify the type of physical activity to effectively manage overweight and obesity. Aerobic exercise namely high intensity interval training have been reported to reduce the body mass, fat%, and waist circumference. Investigators believe that high intensity interval training would help in controlling the various anthropometric variables namely the body mass index, waist circumference, and fat% in trunk region in physically inactive overweight adults.

ELIGIBILITY:
Inclusion Criteria:

* Either gender
* Aged 18-25 years
* Physically Inactive

Exclusion Criteria:

* Any medical condition that restrict the participants to participate in physical exercise
* Blood pressure of more than 140/90 mmHg
* Participants taking any medication that causes drowsiness

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | Change from Baseline Body Mass Index at 4 weeks
Waist Circumference | Change from Baseline Waist Circumference at 4 weeks
Fat Percentage at Trunk Region | Change from Baseline Fat Percentage at Trunk Region at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia